CLINICAL TRIAL: NCT03899610
Title: A Phase II Study of Neoadjuvant Chemotherapy Plus Durvalumab (MEDI4736) and Tremelimumab in Advanced-stage Ovarian Cancer (TRU-D)
Acronym: KGOG3046
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: AstraZeneca (Industry); Samsung Genomic Institute (Unknown); Seoul National University Hospital (Other); Samsung Medical Center (Other); Korean Gynecologic Oncology Group (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0083; KGOG3046 (Other: KGOG); ESR-17-13142 (Other: AstraZeneca)
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV
Keywords: TRU-D
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is single arm phase II study to evaluate efficacy and safety of durvalumab and tremelimumab and chemotherapy in treatment-naïve clinical stage IIIC/IV ovarian cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy+Durvalumab+Tremelimumab (Experimental): 1. Neoadjuvant treatment:
     Standard chemotherapy + Durvalumab + Tremelimumab Durvalumab : 1500mg q3 weeks (total 3 dosing) Tremelimumab : 75mg q 3 weeks (total 3 dosing) Chemotherapy regimen: Paclitaxel 175 mg/m2 , Carboplatin AUC 5-6 q3 weeks (total 3 dosing)
  2. Interval debulking surgery
  3. Adjuvant treatment:
  Standard chemotherapy + Durvalumab Durvalumab; 1120mg q3 weeks (total 12 dosing) Chemotherapy regimen: Paclitaxel 175mg/m2, carboplatin AUC 5-6 q 3weeks (total3 dosing)
  Interventions: Drug: Neoadjuvant chemotherapy+Durvalumab+Tremelimumab

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy+Durvalumab+Tremelimumab — 1. Neoadjuvant treatment:
     Standard chemotherapy + Durvalumab + Tremelimumab Durvalumab : 1500mg q3 weeks (total 3 dosing) Tremelimumab : 75mg q 3 weeks (total 3 dosing) Chemotherapy regimen: Paclitaxel 175 mg/m2 , Carboplatin AUC 5-6 q3 weeks (total 3 dosing)
  2. Interval debulking surgery
  3. Adjuvant treatment:
  Standard chemotherapy + Durvalumab Durvalumab; 1120mg q3 weeks (total 12 dosing) Chemotherapy regimen: Paclitaxel 175mg/m2, carboplatin AUC 5-6 q 3weeks (total3 dosing)

SUMMARY:
The primary objective of this trial is to evaluate the synergistic effects of durvalumab and tremelimumab plus chemotherapy in advanced-stage ovarian cancer.

Ovarian cancer is the deadliest gynecologic cancer. The current standard therapy is surgical cytoreduction followed by taxane-platinum combination chemotherapy. However, most patients with advanced-stage ovarian cancer will experience a relapse of disease. Therefore, there is an urgent need to improve outcomes of patients with this aggressive cancer.

Research hypothesis: Adding durvalumab and tremelimumab to current neoadjuvant chemotherapy (front-line therapy) in advanced-stage ovarian cancer can increase response rate and improve patient's outcome such as progression-free survival and overall survival with minimal effects on safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of ovary, fallopian tube, primary peritoneum
2. Clinical stage IIIC/IV
3. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Female aged 20 years older at the time of acquisition of informed consent
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1
6. Must have life expectancy of at least 16 weeks
7. Body weight >30kg
8. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL) Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Participation in another clinical study with an investigational product during the last 60 days
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Any previous treatment with anti-PD-1, PD-L1, CTLA-4 (including durvalumab and tremelimumab)
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
6. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable. <<amend as required based on any combination studies with other anticancer agents>>
7. Major surgical procedure (except diagnostic laparoscopy) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
11. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1/2 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localised breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than two years prior to registration, and that the patient remains free of recurrent or metastatic disease
12. History of leptomeningeal carcinomatosis
13. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
14. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) << For durvalumab ±tremelimumab in combination with an agent with pro-arrhythmic potential or where effect of the combination on QT is not known if this criterion should be retained. Patient safety and the cardiac EKG should be consulted as needed>>.
15. History of active primary immunodeficiency

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 12 months
  12-months progression-free survival rate will be estimated, and 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Response rate | 9 weeks
  Response rate by RECIST version 1.1 after neoadjuvant chemotherapy(after the completion of 3rd cycle)
Immune-related response | 9 weeks
  Immune-related response after neoadjuvant chemotherapy(after the completion of 3rd cycle)
Response rate by PERCIST | 9 weeks
  Response rate by PERCIST after neoadjuvant chemotherapy(after the completion of 3rd cycle)
R0 rate | at interval debulking surgery after 9 weeks
  R0 rate of IDS(interval debulking surgery) after neoadjuvant chemotherapy(after the completion of 3rd cycle)
The rate of chemotherapy response score 3 | 9 weeks
  The rate of chemotherapy response score 3 after neoadjuvant chemotherapy(after the completion of 3rd cycle)
Overall survival | up to 5 years
  Overall survival up to 5 years
Proportion of patients with grade 3 or more treatment-related adverse events(except hematologic toxicity) graded by CTCAE v5 in neoadjuvant chemotherapy | 9 weeks
  Proportion of patients with grade 3 or more treatment-related adverse events(except hematologic toxicity) graded by CTCAE v5 in neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Korea, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Lee JB, Lim MC, Kim BG, Kim JW, Kim S, Choi CH, Kim HS, Park SY, Lee JY; KGOG investigators. Phase II study of durvalumab and tremelimumab with front-line neoadjuvant chemotherapy in patients with advanced-stage ovarian cancer: primary analysis in the original cohort of KGOG3046/TRU-D. J Immunother Cancer. 2023 Oct;11(10):e007444. doi: 10.1136/jitc-2023-007444. PMID 37865397
- [Derived] Lee JY, Kim JW, Lim MC, Kim S, Kim HS, Choi CH, Yi JY, Park SY, Kim BG; KGOG investigators. A phase II study of neoadjuvant chemotherapy plus durvalumab and tremelimumab in advanced-stage ovarian cancer: a Korean Gynecologic Oncology Group Study (KGOG 3046), TRU-D. J Gynecol Oncol. 2019 Nov;30(6):e112. doi: 10.3802/jgo.2019.30.e112. PMID 31576697